CLINICAL TRIAL: NCT05679154
Title: Implementation of the Care Process Model for Pediatric Traumatic Stress in Rural Child Advocacy Centers: A Pilot Test of Team-focused Implementation
Brief Title: Team-Focused Implementation in Child Advocacy Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Elizabeth McGuier, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY21010070; K23MH123729 (NIH)
Record Dates: First submitted 2022-12-15; First posted 2023-01-10 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Mental Health Issue; Teamwork
Keywords: Mental health screening; Implementation; Teamwork

STUDY DESIGN:
Intervention Model Description: The trial includes two groups: team-focused implementation and standard implementation (comparison group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Team-focused Implementation (Experimental)
  Interventions: Behavioral: Team-focused Implementation
- Standard Implementation (Active Comparator)
  Interventions: Behavioral: Standard Implementation

INTERVENTIONS:
Behavioral: Team-focused Implementation — CACs randomized to the experimental condition (n = 2) will participate in team-focused implementation. They will receive team development interventions (e.g., goal-setting exercise, training in communication skills) integrated with standard CPM-PTS training and technical assistance strategies.
  Arms: Team-focused Implementation
Behavioral: Standard Implementation — CACs randomized to the comparison condition (n = 2) will receive standard training and technical assistance strategies to support CPM-PTS implementation. They will receive CPM-PTS materials (e.g., manual, REDCap surveys, referral protocols), an interactive training, and six months of technical assistance.
  Arms: Standard Implementation

SUMMARY:
Child Advocacy Centers (CACs) are well-positioned to identify children at risk for mental health problems and to facilitate access to evidence-based treatments. Implementation of standardized mental health screening and referral protocols may improve recognition of mental health needs and facilitate treatment engagement. Implementation strategies that improve teamwork may enhance implementation outcomes in team-based settings like CACs. In this study, CACs will implement the Care Process Model for Pediatric Traumatic Stress (CPM-PTS) and be randomized to either team-focused implementation or standard implementation. The study aims are to evaluate the feasibility of team-focused implementation and the effect of the CPM-PTS on caregiver understanding of mental health needs and intentions to initiate treatment.

DETAILED DESCRIPTION:
This study is a pilot cluster randomized controlled hybrid Type II effectiveness-implementation trial in 4 rural Child Advocacy Centers. All CACs will implement the Care Process Model for Pediatric Traumatic Stress (CPM-PTS), a mental health screening and referral protocol. CACs will be randomized to team-focused implementation (n = 2) or standard implementation (n = 2). The study is designed to evaluate the acceptability, appropriateness, and feasibility of team-focused implementation strategies. It will also test the effect of the CPM-PTS on caregiver understanding of mental health needs and intentions to initiate treatment. Mixed methods will be used to evaluate the feasibility of team-focused implementation, test the effect of team strategies on teamwork, and assess implementation outcomes. Administrative data collected anonymously from caregivers will be used to test the effectiveness of the CPM-PTS.

ELIGIBILITY:
Inclusion Criteria:

* Individuals at least 18 years of age who are members of the multidisciplinary team at the participating CACs.

Exclusion Criteria:

* Under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Acceptability of team-focused implementation assessed by the Acceptability of Intervention Measure | Baseline
  Perceived acceptability of team-focused implementation will be assessed with items from the Acceptability of Intervention Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions (range 1-5).
Acceptability of team-focused implementation assessed by the Acceptability of Intervention Measure | Month 6
  Perceived acceptability of team-focused implementation will be assessed with items from the Acceptability of Intervention Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions (range 1-5).
Acceptability of team-focused implementation assessed by the Acceptability of Intervention Measure | Month 12
  Perceived acceptability of team-focused implementation will be assessed with items from the Acceptability of Intervention Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions (range 1-5).
Appropriateness of team-focused implementation assessed by the Intervention Appropriateness Measure | Baseline
  Perceived appropriateness of team-focused implementation will be assessed with items from the Intervention Appropriateness Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions (range 1-5).
Appropriateness of team-focused implementation assessed by the Intervention Appropriateness Measure | Month 6
  Perceived appropriateness of team-focused implementation will be assessed with items from the Intervention Appropriateness Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions (range 1-5).
Appropriateness of team-focused implementation assessed by the Intervention Appropriateness Measure | Month 12
  Perceived appropriateness of team-focused implementation will be assessed with items from the Intervention Appropriateness Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions (range 1-5).
Feasibility of team-focused implementation assessed by the Feasibility of Intervention Measure | Baseline
  Perceived feasibility of team-focused implementation will be assessed with items from the Feasibility of Intervention Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions (range 1-5).
Feasibility of team-focused implementation assessed by the Feasibility of Intervention Measure | Month 6
  Perceived feasibility of team-focused implementation will be assessed with items from the Feasibility of Intervention Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions (range 1-5).
Feasibility of team-focused implementation assessed by the Feasibility of Intervention Measure | Month 12
  Perceived feasibility of team-focused implementation will be assessed with items from the Feasibility of Intervention Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions (range 1-5).

SECONDARY OUTCOMES:
Change in team functioning from baseline to 6-month follow-up | Baseline, month 6
  Affective, behavioral, and cognitive processes and states will be assessed with survey items rated on Likert scales. Scores will be averaged; higher scores indicate more adaptive team functioning (range 1-7).
Change in team functioning from baseline to 12-month follow-up | Baseline, month 12
  Affective, behavioral, and cognitive processes and states will be assessed with survey items rated on Likert scales. Scores will be averaged; higher scores indicate more adaptive team functioning (range 1-7).
Change in team performance from baseline to 6- and 12-month follow-up | Baseline, month 6, month 12
  The overall quality of work done by the team will be assessed with Edmondson's (1999) Team Performance scale (5 items rated on a 7-point Likert scale). Scores will be averaged; higher scores indicate better performance (range 1-7).
CPM-PTS Acceptability assessed by the Acceptability of Intervention Measure | Month 6
  Perceived acceptability of the CPM-PTS will be assessed with items from the Acceptability of Intervention Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions (range 1-5).
CPM-PTS Acceptability assessed by the Acceptability of Intervention Measure | Month 12
  Perceived acceptability of the CPM-PTS will be assessed with items from the Acceptability of Intervention Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions (range 1-5).
CPM-PTS Appropriateness assessed by the Intervention Appropriateness Measure | Month 6
  Perceived appropriateness of the CPM-PTS will be assessed with items from the Intervention Appropriateness Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions (range 1-5).
CPM-PTS Appropriateness assessed by the Intervention Appropriateness Measure | Month 12
  Perceived appropriateness of the CPM-PTS will be assessed with items from the Intervention Appropriateness Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions (range 1-5).
CPM-PTS Feasibility assessed by the Feasibility of Intervention Measure | Month 6
  Perceived feasibility of the CPM-PTS will be assessed with items from the Feasibility of Intervention Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions (range 1-5).
CPM-PTS Feasibility assessed by the Feasibility of Intervention Measure | Month 12
  Perceived feasibility of the CPM-PTS will be assessed with items from the Feasibility of Intervention Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions (range 1-5).
CPM-PTS Adoption | From start of the study for up to 12 months after CPM-PTS implementation
  Adoption will be indicated by the number of days from training to the first completed screening.
CPM-PTS Reach | Monthly for 12 months after CPM-PTS implementation
  Reach will be indicated by screening rates (i.e., completed screenings / eligible children) and calculated for monthly and quarterly periods (possible range 0-100%).

OTHER OUTCOMES:
Caregiver understanding of child mental health needs | Collected immediately after CAC visit for all caregivers served during an 18 month period (beginning 6 months before CPM-PTS implementation and continuing for 12 months after implementation)
  Caregivers will rate 1 item assessing their understanding of their child's mental health needs on a 4-point Likert scale (range 1-4) in an anonymous end of visit survey.
Caregiver intention to initiate mental health services | Collected immediately after CAC visit for all caregivers served during an 18 month period (beginning 6 months before CPM-PTS implementation and continuing for 12 months after implementation)
  Caregivers will rate 1 item assessing their intention to initiate mental health services for their child on a 5-point Likert scale (range 1-5) in an anonymous end of visit survey.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth McGuier, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available upon reasonable request as allowed by IRB regulations and after manuscripts reporting the main findings are accepted for publication.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after manuscripts reporting the main findings are accepted for publication.
Access Criteria: Contact the principal investigator to request access to the deidentified data.

REFERENCES:
- [Derived] McGuier EA, Aarons GA, Wright JD, Fortney JC, Powell BJ, Rothenberger SD, Weingart LR, Miller E, Kolko DJ. Team-focused implementation strategies to improve implementation of mental health screening and referral in rural Children's Advocacy Centers: study protocol for a pilot cluster randomized hybrid type 2 trial. Implement Sci Commun. 2023 May 26;4(1):58. doi: 10.1186/s43058-023-00437-z. PMID 37237302